CLINICAL TRIAL: NCT01996163
Title: The Effect of Gender on the Consumption of Pain Medication in Infants Undergoing Craniosynostosis Repair or Untethering of Cord in ITU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-13-FS-0561-13-CTIL
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Craniosynostosis Repair; Untethering of Cord

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Male
- Female

SUMMARY:
Postoperative pain is a major concern in routine management of children admitted to pediatric intensive care treatment. There are significant negative physiological and psychological ramifications of postoperative pain such as impairment of cardiac function due to tachycardia, restlessness in an intubated patient requiring increase dosage of sedative and paralytic drugs and reduced patient cooperation in the healing process.

The main body of evidence dealing with gender differences in pain perception and treatment stems from studies in the adult and adolescent population as the gonadal hormones have a central role in the way one experiences pain The hypothesis of this study is that there is a difference in the perception of pain, the amount of analgesia used and the response to pain medication between male and female infants undergoing craniosynostosis repair or untethering of cord.

ELIGIBILITY:
Inclusion Criteria:

All infants 0-1 year old, admitted to PICU after craniosynostosis repair or untethering of cord.

Exclusion Criteria:

1. Contraindication to analgesic medication
2. Infants with neurologic deficits that may hinder the assessment of pain severity such as facial nerve palsy and limb paralysis.
3. Ventilated infants.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants 0-1 year old, admitted to PICU after craniosynostosis repair or untethering of cord.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The average amount per kg of analgesic medications in male and female infants 0-1 year old. | The first 24h after surgery
The average reduction in pain severity score after receiving analgesics in male and female infants. | 24h after surgery